CLINICAL TRIAL: NCT04554264
Title: Complicated Grief in ICU in the Aftermath of COVID-19
Acronym: DEPARTS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: University Hospital, Lille (Other); University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PI2020_843_0071
Record Dates: First submitted 2020-09-02; First posted 2020-09-18 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Complicated Grief; Intensive Care; Covid19
Keywords: Complicated grief; Intensive Care; Covid19
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — Inventory of Complicate Grief (ICG) score in relative from patients who died in ICU after SARS-Cov2 infection. This is the most commonly used assessment tool for complicated grief which focuses on different symptoms than depression or anxiety. A score > 25 indicate complicated grief.

SUMMARY:
An increased proportion of deaths occur in the intensive care unit (ICU). Some amenable factors such as end-of-life practices may contribute to complicated grief.

Because of the COVID-19 pandemic, visitor restrictions in health care facilities have been implemented. Families were also unable to implement usual funerals. The investigators hypothesize that these policies and practices may impact grief during covid-19 pandemic. The aim of this study is to evaluate the prevalence of complicated grief after death of a relative in the ICU during the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* adult relative (>18 years)
* adult relative from patients who died in ICU after SARS-COV-2 infection

Exclusion Criteria:

* adult relative (<18 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Proportion of complicated grief 4 month after death in relative from patients who died in ICU after covid-19 infection evaluate with ICG score. | 4 months after relative death
  Proportion of complicated grief 4 month after death in relative from patients who died in ICU after covid-19 infection evaluate with ICG score.
  The primary outcome measure is the Inventory of Complicate Grief (ICG) score. This is the most commonly used assessment tool for complicated grief which focuses on different symptoms than depression or anxiety. A score > 25 indicate complicated grief.
  All patients who died in ICU after SARS-Cov-2 infection will be identify. Their relatives (spouse, children and relative who served as a surrogate) will also be identify. Relatives will be included up to 4 months after the time of death.
Proportion of complicated grief 6 month after death in relative from patients who died in ICU after covid-19 infection evaluate with ICG score. | 6 months after relative covid-19 death
  Proportion of complicated grief 6 month after death in relative from patients who died in ICU after covid-19 infection evaluate with ICG score.
  The primary outcome measure is the Inventory of Complicate Grief (ICG) score. This is the most commonly used assessment tool for complicated grief which focuses on different symptoms than depression or anxiety. A score > 25 indicate complicated grief.
  All patients who died in ICU after SARS-Cov-2 infection will be identify. Their relatives (spouse, children and relative who served as a surrogate) will also be identify. Relatives will be included up to 6 months after the time of death.
Proportion of complicated grief 12 month after death in relative from patients who died in ICU after covid-19 infection evaluate with ICG score. | 12 months after relative covid-19 death
  Proportion of complicated grief 12 month after death in relative from patients who died in ICU after covid-19 infection evaluate with ICG score.
  The primary outcome measure is the Inventory of Complicate Grief (ICG) score. This is the most commonly used assessment tool for complicated grief which focuses on different symptoms than depression or anxiety. A score > 25 indicate complicated grief.
  All patients who died in ICU after SARS-Cov-2 infection will be identify. Their relatives (spouse, children and relative who served as a surrogate) will also be identify. Relatives will be included up to 12 months after the time of death.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No